CLINICAL TRIAL: NCT05387616
Title: A Prospective Multicenter Phase 2 Study of the Chemotherapy-Free Combination of the Intravenous Phosphatidylinositol-3-Kinase (PI3K) Inhibitor Copanlisib in Combination With Obinutuzumab in Patients With Previously Untreated Follicular Lymphoma (FL) and a High Tumor Burden
Acronym: Alternative-C
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Roche Pharma AG (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Christian Schmidt, MD, Dr. Christian Schmidt, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alternative-C; 2018-004038-13 (EudraCT Number)
Record Dates: First submitted 2022-01-27; First posted 2022-05-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — copanlisib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Copanlisib + Obinutuzumab (Experimental)
  Interventions: Drug: Copanlisib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Copanlisib — Induction therapy will comprise 6 cycles of copanlisib, administered by intravenous Infusion at a dose of 60 mg on day 1,8,15 of cycles 1-6 to be given every 28 days.
  Consolidation therapy will comprise another 24 weeks of copanlisib in patients with clinical Remission 28 days after the last induction cycle. It will be administered by intravenous Infusion at a dose of 60 mg on days 1 and 15 of cycles 7 - 12 to be given every 28 days.
  Maintenance therapy will comprise another 72 weeks of copanlisib in patients with clinical remissions 28 days after the last consolidation cycle.
  Other Names: ALIQOPA™
Drug: Obinutuzumab — Induction therapy will comprise 6 cycles of obinutuzumab, administered by intravenous infusion at a dose of 1000 mg on days 1,8, 15 of cycle 1 and on day 1 of cycles 2 - 6 to be given every 28 days.
  Consolidation therapy will comprise of another 24 weeks of obinutuzumab in patients with clinical remission 28 days after the last induction cycle. Obinutuzumab will be applied at a dose of 1000 mg by intravenous infusion every 8 weeks.
  Maintenance therapy will comprise another 72 weeks in patients with clinical remission 28 days after the last consolidation cycle. Obinutuzumab will be applied at a dose of 1000 mg by intravenous infusion every 8 weeks.
  Other Names: GAZYVARO®

SUMMARY:
The Alternative-C Trial is a prospective, multicenter Phase 2 Study to evaluate the efficacy of the chemotherapy-free combination of copanlisib and obinutuzumab in patients with previously untreated follicular lymphoma (FL) and a high tumor burden. Additionally, the combination should be evaluated in terms of secondary efficacy endpoints, treatment compliance, safety and patient-reported symptoms. The study Population includes Patients > 18 years of age with histologically confirmed follicular lymphoma grade 1, 2 or 3A with Ann Arbor Stage III/IV or stage II not suitable for radiotherapy and in need of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be included in the study, if they meet all of the following criteria:
* Histologically confirmed follicular lymphoma grade 1, 2 or 3A with a biopsy performed within 12 months before study entry and with material available for central review and complementary scientific analyses
* Ann Arbor stage III/IV, or stage II not suitable for radiotherapy, or stage II bulky disease
* Age ≥ 18 years
* No prior lymphoma therapy
* Need for start of therapy as defined by at least one of the following criteria:

  * bulky disease at study entry according to the GELF criteria (nodal or extranodal mass > 7 cm in its greatest diameter)
  * B symptoms (fever, drenching night sweats, or unintentional weight loss of > 10% of normal body weight over a period of 6 months or less)
  * hematopoietic insufficiency (granulocytopenia < 1500/µl, Hb < 10 g/dl, thrombocytopenia < 100000/µl)
  * compressive syndrome or high risk for compression syndrome
  * pleural/peritoneal effusion
  * symptomatic extranodal manifestations
* At least one bi-dimensionally measurable lesion (> 2 cm in its largest dimension by CT scan or MRI)
* Performance status ≤ 2 on the ECOG scale
* Adequate hematologic function (unless abnormalities are related to NHL), defined as follows:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1500/µl
  * Platelet count ≥ 75000/µl
* Women are not breast feeding, are using highly effective contraception (see section 11.4.1), are not pregnant, and agree not to become pregnant during participation in the study and during the 18 months thereafter (pregnancy testing is mandatory for premenopausal women).
* Men agree not to father a child during participation in the study and during the 18 months thereafter.
* Written informed consent

Exclusion criteria:

Subjects will not be included in the study if any of the following criteria apply:

* Transformation to high-grade lymphoma (secondary to "low grade" FL)
* Grade 3B follicular lymphoma
* Presence or history of CNS disease (either CNS lymphoma or leptomeningeal lymphoma)
* Known hypersensitivity to any of the study drugs
* Known sensitivity to murine products
* Patients with HbA1c > 8.5 % at Screening
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's assessment)
* Regular use of corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 20 mg/day prednisone or administered as prephase treatment according to study protocol (see section 7.2 of study protocol)
* Concomitant use of strong CYP3A4 inhibitors and/or inducers
* Prior or concomitant malignancies except:

  * non-melanoma skin cancer or adequately treated in carcinoma in situ of the cervix
  * other malignant diseases not specified above which have been curatively treated by surgery alone and from which subject is disease-free for ≥ 5 years without further treatment
* Serious disease interfering with a regular therapy according to the study protocol:

  * Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
  * pulmonary (e.g. chronic lung disease with hypoxemia)
  * endocrine (e.g. severe, not sufficiently controlled diabetes mellitus)
  * renal insufficiency (unless caused by the lymphoma): creatinine > 2x normal value and/or creatinine clearance < 50 ml/min)
  * impairment of liver function (unless caused by the lymphoma): transaminases > 3x normal or bilirubin > 2.0 mg/dl (unless caused by known Morbus Meulengracht [Gilbert-Meulengracht-Syndrome])
* Positive test results for chronic HBV infection (defined as positive HBsAg serology) Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing.

Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible.

* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing) Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
* Known history of HIV seropositive status
* Patients with a history of confirmed PML
* Vaccination with a live vaccine within 28 days prior to registration
* Recent major surgery (within 4 weeks prior to the start of Cycle 1)
* History of stroke or intracranial hemorrhage within 6 months prior to registration
* Serious underlying medical conditions, which could impair the ability of the patient to undergo the treatment offered in the study (e.g. ongoing infection, gastric ulcers, active autoimmune disease)
* Treatment within another clinical study within 30 days prior to study entry
* Prior organ, bone marrow, or peripheral blood stem cell transplantation
* Known or persistent abuse of medication, drugs, or alcohol
* Any other co-existing medical or psychological condition that will preclude participation in the study or compromise ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
One-year progression-free survival (PFS) probability from study registration | 1 year
  The rate of patients achieving a progression free survival of more than one year after registration (one-year PFS rate) will serve as early readout for efficacy.

SECONDARY OUTCOMES:
Complete remission (CR) rates and overall response (CR or partial remission, PR) rates | at end of induction (month 6), at end of consolidation (month 12), and at end of maintenance (month 30)
Progression free survival from registration | continuous observation up to 78 months
Duration of response | from end of induction to progression or death assessed up to 72 months
Cumulative incidence of progression | from registration to end of study assessed up to 78 months
Failure-free survival | from start of therapy assessed up to 78 months
  event defined by failure to achieve a CR/PR after 6 months or progression after CR or PR or death from any cause
Time to next anti-lymphoma therapy and time to next chemotherapy based treatment | from start of first-line therapy up to 78 months
Overall survival | from registration up to 78 months
Treatment associated adverse events | continuous observation up to 78 months
Percentage of MRD-negative patients | therapy (month 12), and at end maintenance therapy (month 30)
Duration of molecular remission for MRD negative patients | from end of induction therapy up to 72 months
Cumulative incidence of secondary transformations to aggressive lymphoma | ongoing observation up to 78 months
Cumulative incidence of secondary malignancies | ongoing observation up to 78 months
Percentage of patients with compliance to therapy | after 6, 12, and 30 months
Frequency of patient-reported lymphoma symptoms and concerns (FACT-Lym) | Baseline, End of Induction, End of Consolidation, End of Maintenance, and every 6 months during FU for at least 2 years until end of the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmidt, Dr., Principal Investigator — LMU Klinikum, Medical department III
Locations (40):
- Germany (40):
  - LMU Klinikum, München, Bavaria
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum am Urban, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Cancer Center Dachau, Dachau
  - Städtisches Klinikum Dessau, Dessau
  - Gemeinschaftspraxis Dr. med. J. Mohm und Dr. med. G. Prange-Krex, Dresden
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Praxis für Hämatologie und Onkologie, Koblenz
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - Universitätsklinik Mannheim, Mannheim
  - Kliniken Maria Hilf GmbH, Krankenhaus St. Franziskus, Mönchengladbach
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Klinikum rechts der Isar der TU München, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Universitätsklinikum Münster, Münster
  - Friedrich Ebert Krankenhaus, Neumünster
  - Rheinland Klinikum, Lukaskrankenhaus Neuss, Neuss
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsmedizin Rostock, Rostock
  - Klinikum Südstadt Rostock, Rostock
  - Gemeinschaftspraxis Dr. med. G.A. Jacobs, Saarbrücken
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Petrus Kankenhaus, Wuppertal
  - Hämatologisch-Onkologische Schwerpunktpraxis, Würzburg

IPD SHARING:
Plan to Share IPD: No